CLINICAL TRIAL: NCT04538274
Title: A Peer-driven Intervention to Help Patients Resume CPAP Therapy Following Discontinuation: a Multicenter, Randomized Clinical Trial with Patient Involvement
Brief Title: Trained Patient Involvement to Promote the Resumption of CPAP in Patients Who Have Discontinued Its Use
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-06; NCT04774692 (obsolete NCT alias)
Record Dates: First submitted 2020-08-14; First posted 2020-09-04 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Sleep Apnea; CPAP adherence; Patient and Public Involvement (PPI); cognitive-behavioural and motivation enhancement therapies; Patient Involvement (PI)
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Patient Participation

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicentre, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient researcher intervention (Experimental): Intervention conducted by trained patient researchers to restart CPAP in addition to usual care
  Interventions: Behavioral: peer-driven intervention
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: peer-driven intervention — Trained patient researchers will conduct 3 motivational sessions, according to the principle of motivational enhancement and cognitive-behavioral therapies, by videoconference meetings of 45 to 60 minutes duration with 5 to 8 patients within 6 months after each patient's inclusion.
  Arms: Patient researcher intervention

SUMMARY:
The primary objective of this randomized clinical trial is to evaluate the role of patient researchers in promoting the resumption of CPAP therapy in apneic patients who had previously stopped CPAP

DETAILED DESCRIPTION:
Obstructive Sleep Apnoea syndrome (OSA) is one of the most frequent chronic disease presenting with or without symptoms of excessive daytime sleepiness (EDS) and being accompanied by neurocognitive, cardiovascular and metabolic complications.

The first line therapy of obstructive sleep apnoea is continuous positive airway pressure (CPAP). CPAP is highly effective in symptomatic patients for reducing EDS and improving daily functioning, cognitive function, mood and quality of life. However, success of CPAP treatment is hampered by long term nonadherence in nearly half of patients. Non adherence to CPAP is less and less related to technical problems, but rather to users' profile, their representations of OSA and the benefits experienced from CPAP. Cognitive-behavioural and motivation enhancement therapies can promote adherence to CPAP treatment. In addition to health professionals, patients and public involvement (PPI) is more and more advocated in the field of education and research. Nevertheless, the level of evidence regarding efficacy of PPI and patient researchers remains to be demonstrated. The aim of this randomized clinical trial is to evaluate the role of patient researchers in promoting the resumption of CPAP therapy in apneic patients who had previously stopped CPAP

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Diagnosed with of severe OSA (AHI ≥ 30 events/hour)
* Discontinuation of CPAP 4 to 12 months after initiation Followed by the home health care provider Agiradom
* Access to a computer and/or tablet and an internet connection
* Oral and written French
* Able to provide written informed consent
* Affiliated to social security or beneficiary of such a scheme

Exclusion Criteria:

* CPAP cessation due to a resolution of the OSAS (e.g. weight loss after bariatric surgery) or another pathology that prevents the continuation of treatment (e.g. ENT surgery, etc.).
* Severe and/or unstable comorbidity that required hospitalisation for decompensation in the previous year (heart, kidney, respiratory, liver, psychiatric or other insufficiency).
* Patient being treated with a mandibular advancement orthosis
* Lack of availability (e.g. night worker or patient who travels frequently, etc.).
* Current participation in, participation in the month prior to inclusion in another clinical intervention research study that may impact the study: this impact is left to the investigator's discretion.
* Referred to in Articles L1121-5 to L1121-8 of the CSP (corresponds to all protected persons: pregnant woman, breastfeeding mother, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-02-18 (Estimated); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact of a 6-month, peer-driven intervention to promote the resumption of CPAP after discontinuation | 6 months after inclusion
  The range of patients reusing CPAP in the intervention group The difference in percentages of patients who reuse CPAP between the peer-driven intervention group and the control group.

SECONDARY OUTCOMES:
Evaluate the impact of the peer-driven intervention on adherence to CPAP compared to the control group | 6 month after inclusion
  the difference in CPAP compliance (average hours of use/night) between the AP intervention group and a control group
Evaluate the impact of the peer-driven intervention on adherence to CPAP compared to the control group | 6 month after inclusion
  the difference in percentages of patients who reuse to CPAP with at least 4 hours' use /night for 70% of nights
Disease-specific quality of life | At inclusion and after 6 months
  The Functional Outcomes of Sleep Questionnaire (FOSQ10) will be completed at inclusion (M0) and at the 6-month follow-up (M6).
  This variable will be used to assess predictors of positive response to patient researcher intervention
Patient Self-Efficacy Measure for Sleep Apnea | At inclusion and after 6 months
  The Self-Efficacy Measure for Sleep Apnea (SEMSA) questionnaire, a tool with strong psychometric properties and with the potential for identifying patient perceptions will be completed at inclusion (M0) and at the 6-month follow-up (M6). This variable will be used to assess predictors of positive response to patient researcher intervention
Patient knowledge, skill, and confidence for self-management | At inclusion and after 6 months
  The Patient Activation Measure (PAM) qestionnaire, a measure that assesses patient knowledge, skill, and confidence for self-management, will be completed at inclusion (M0) and at the 6-month follow-up (M6) This variable will be used to assess predictors of positive response to patient researcher intervention
Patient satisfaction and peer satisfaction | At 6 month after inclusion
  Patient satisfaction with the peer-driven intervention at 6 months will be measured on a 4-point Likert scale : very dissatisfied, dissatisfied, satisfied, very satisfied.
  Satisfaction of PI representatives will be measured on a 4-point Likert scale: very dissatisfied, dissatisfied, satisfied, very satisfied.
Feasibility and the execution of the peer-driven intervention | At 6 month after inclusion
  Evaluate the feasibility and the execution of the peer-driven intervention
Age | inclusion
  This variable will be used to assess predictors of positive response to patient researcher intervention
Gender | inclusion
  This variable will be used to assess predictors of positive response to patient researcher intervention
BMI Body Mass Index | inclusion
  This variable will be used to assess predictors of positive response to patient researcher intervention
marital status with infants (<10 years) or not | inclusion
  This variable will be used to assess predictors of positive response to patient researcher intervention
Education level | inclusion
  This variable will be used to assess predictors of positive response to patient researcher intervention
employment and socio-professional status | inclusion
  This variable will be used to assess predictors of positive response to patient researcher intervention
alcohol-smoking status | inclusion
  This variable will be used to assess predictors of positive response to patient researcher intervention
fragility and social precariousness | inclusion
  EPICES score will be used to assess predictors of positive response to patient researcher intervention
medication adherence | inclusion
  Girerd Score. This variable will be used to assess predictors of positive response to patient researcher intervention
OSA history | inclusion
  date of diagnosis of OSA
CPAP treatment | inclusion
  Date of initiation of CPAP and date and cause of CPAP discontinuation
Baseline Apnea-Hypopnea Index (AHI) | inclusion
  This variable will be used to assess predictors of positive response to patient researcher intervention
Excessive daytime sleepiness (EDS score) | inclusion
  Epworth Sleepiness Scale will be used to assess predictors of positive response to patient researcher intervention
Comorbidities | inclusion
  Charlson index will be used to assess predictors of positive response to patient researcher intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merle R, Pison C, Logerot S, Deschaux C, Arnol N, Roustit M, Tamisier R, Pepin JL, Borel JC. Peer-driven intervention to help patients resume CPAP therapy following discontinuation: a multicentre, randomised clinical trial with patient involvement. BMJ Open. 2021 Oct 14;11(10):e053996. doi: 10.1136/bmjopen-2021-053996. PMID 34649850